CLINICAL TRIAL: NCT01957527
Title: Offset of Ticagrelor's Effect on Endothelial Function as Assessed With Peripheral Arterial Tonometry (EndoPAT Assay)
Status: Completed | Type: Observational
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Other Study IDs: PATRASCARDIOLOGY-15
Record Dates: First submitted 2013-09-30; First posted 2013-10-08 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Artery Disease; Endothelial Function
Keywords: ticagrelor; endothelial function; peripheral arterial tonometry
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ticagrelor discontinuation
  Interventions: Device: Peripheral arterial tonometry (EndoPAT)

INTERVENTIONS:
Device: Peripheral arterial tonometry (EndoPAT)

SUMMARY:
Ticagrelor administration, whose molecule resembles to adenosine, led to reduction in overall mortality and thrombotic cardiovascular (CV) events when directly compared to clopidogrel in the PLATO trial, implicating possible pleiotropic actions for the drug. It has been shown that ticagrelor increases adenosine concentration, by interfering with its red blood cells' uptake and by inducing the release of ATP which is then converted to adenosine. Recent studies in healthy volunteers and patients with coronary artery disease (CAD) have shown that ticagrelor increases the coronary blood flow in response to intravenous adenosine administration. Ticagrelor administration, in comparison with other P2Y12 inhibitors, may influence the endothelial function, as assessed by the Peripheral Arterial Tonometry method (EndoPAT 2000 system (Itamar Medical, Caesarea, Israel), which is a method for evaluating endothelial dysfunction and has been found to positively correlate with flow mediated dilatation (FMD).

This is a prospective, observational study, which will be conducted in patients with coronary artery disease subjected to percutaneous coronary intervention (PCI) under ticagrelor maintenance dose (MD) 90mg x 2, who are about to stop treatment, due to completion of 1 year antiplatelet therapy. Eligible patients will be subjected to peripheral arterial tonometry at Day 0 (immediately after receiving the last pill of ticagrelor) and at day 2 and day 5 post study drug discontinuation. Peripheral blood sample will be taken from the patients at Day 0 for genotype analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18-80 years old
2. Patients with Coronary Artery Disease receiving ticagrelor maintenance dose (MD) 90mg x 2 and are about to discontinue the treatment due to the completion of 1 year of dual antiplatelet therapy.
3. Patients giving written Informed Consent.

Exclusion Criteria:

1. Acute Coronary Syndrome
2. Foreseeable need for anticoagulant treatment within the next 5 days
3. Severe non-regulated with theophylline/aminophylline administration chronic obstructive pulmonary disease
4. Creatinine Clearance <30ml/min/1.73mm2
5. HbA1c > 10mg/dl

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease under ticagrelor maintenance dose, who are about to discontinue ticagrelor, due to completion of 12 months dual antiplatelet therapy.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Reactive Hyperemia Index (RHI) on Day 0 and on Day 5 | 5 days
  Reactive Hyperemia Index (RHI) on Day 0 will be compared to RHI on Day 5

SECONDARY OUTCOMES:
Reactive Hyperemia Index (RHI) on Day 0 and on Day 2 | 2 days
  Reactive Hyperemia Index (RHI) on Day 0 will be compared to RHI on Day 2
Reactive Hyperemia Index (RHI) on Day 2 and on Day 5 | 3 days
  Reactive Hyperemia Index (RHI) on Day 2 will be compared to RHI on Day 5
The percentage of patients with RHI<1.67 on Day 0 and on Day 5 | 5 days
The percentage of the patients with RHI<1.67 on Day 0 and on Day 2 | 2 days
The percentage of the patients with RHI<1.67 on Day 2 and on Day 5 | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Patras University Hospital, Pátrai, Achaia, Greece